CLINICAL TRIAL: NCT04356872
Title: A Single Arm, Multi Centers, Phase II Study of Sintilimab, Doxorubicin and Ifosfamide at First-line Treatment of Soft Tissue Sarcoma Including Undifferentiated Pleomorphic Sarcoma, Synovial Sarcoma, Myxoid Liposarcoma and De-differentiated Liposarcoma
Brief Title: The Combination of Sintilimab and AI (Doxorubicin, ADM/Ifosfamide, IFO) for the First Line Treatment of Select Type of Metastatic/Unresectable Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Tongji Hospital (Other); Xijing Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Chief Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAIS
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Sarcoma, Soft Tissue
Keywords: PD-1; doxorubicin; ifosfamide; first line treatment
MeSH Terms: conditions — Sarcoma | interventions — sintilimab; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): The patients with metastatic and unresectable soft tissue sarcoma including undifferentiated pleomorphic sarcoma, synovial sarcoma, de-differentiated liposarcoma and myxoid liposarcoma will be enrolled and given sintilimab (PD-1) , doxorubicin and doxorubicin every three weeks for 6 cycles followed by sintilimab mono therapy till disease progression. The first enrolled six patients is safety run-in step for observing drug-limiting toxicity (DLTs). If the combinatory treatment is intolerable, the doses of chemo regimens will be reduced according to drug instruction.
  Interventions: Drug: Sintilimab; Drug: Doxorubicin Hydrochloride; Drug: Ifosfamide

INTERVENTIONS:
Drug: Sintilimab — immune check point inhibitor, 200mg, iv, d1
Drug: Doxorubicin Hydrochloride — ADM, 60mg/m2, iv, d1
  Other Names: ADM
Drug: Ifosfamide — IFO, 1.8 g/m2/d, d1-5
  Other Names: IFO

SUMMARY:
This is a phase II trial to explore the feasibility of PD-1 immune check point inhibitor, sintilimab, in combination of stand of care chemotherapy in first-line treatment of selected soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 years;
* Provide written informed consent;
* Local advanced or metastatic unresectable sarcoma;
* Histologically confirmed undifferentiated pleomorphic sarcoma, synovial sarcoma, de-differentiated liposarcoma and myxoid liposarcoma;
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale;
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
* Life span expectation over 3 months
* Absolute neutrophil count (ANC) ≥1,500/mcL (within 7 days of treatment initiation) ；
* Hemoglobin ≥9 g/dL (within 7 days of treatment initiation) ；
* Platelets ≥ 90,000/mcL (within 7 days of treatment initiation) ；
* Serum creatinine ≤ 1.5 X upper limit of normal (ULN) or creatinine clearance [CrCl]) ≥ 50 mL/min for subject with creatinine levels (within 7 days of treatment initiation) ；
* Serum total bilirubin ≤ 1.5 X ULN (within 7 days of treatment initiation) ；
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 X ULN or =< 5 X ULN for subjects with liver metastases (within 7 days of treatment initiation)；

Exclusion Criteria:

* Prior systemic therapy for advanced and metastatic disease, except adjuvant treatment（not received anthracycline）replase over 6 months;
* Received any testing anti-cancer drugs within four weeks of treatment initiation;
* Prior immune related therapy including but not limited to PD-1, PD-L1, CD137, CTLA4, T cell stimulation, check point inhibitor etc;
* Symptomatic, untreated, or uncontrolled brain metastases present
* clinical meaningful active bleeding;
* Other malignant cancer history rather than soft tissue sarcoma within five year prior to treatment initiation;
* Have active infections requiring therapy;
* Have active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients that require inhaled steroids or local steroid injections would not be excluded from the study. Patients with hypothyroidism not from autoimmune disease that is stable on hormone replacement will not be excluded from the study.
* Pregnant or breast-feeding；
* Any serious or unstable medical condition or mental illness；
* Serious systemic diseases such as heart disease, history of (non-infectious) pneumonitis;
* Active HBV （>10000 copy/ml） and HCV （RNA> 1000copy/ml） infection；
* Positive human immunodeficiency virus (HIV）or any acquired immunodeficiency syndrome, organ implantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate, ORR | up to two years
  the best response rate

SECONDARY OUTCOMES:
progression free survival, PFS | up to three years
  from first dose treatment to disease progression
adverse events, AE | up to three years
  treatment related adverse events, TRAEs
overall survival, OS | up to three years
  overall survival

OTHER OUTCOMES:
PD-L1 expression | up to two years
  PD-L1 expression will be detected by Immunohistologic chemistry, IHC or PCR method
tumor infiltrating lymphocytes measurement | up to two years
  tumor infiltrating lymphocytes will be measured by flowcytometry using tissue and/or peripheral blood sample；

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
not yet decide, need to discuss with all collaborators